CLINICAL TRIAL: NCT02134951
Title: Biomarker Assessment of Glutamatergic Target Engagement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marlene Carlson, Manager, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6925; HHS-N-271-2012-0000-7-I (Other: NIH/NIMH contract number)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Healthy Controls
MeSH Terms: interventions — Ketamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketamine (Experimental): IV infusion of ketamine 0.23mg/kg bolus over 1 minutes followed by 0.58 mg/kg/hr over 30 minutes then 0.29mg/kg/hr over 64 minutes
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Placebo group will receive normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — intravenous infusion of saline solution with ketamine
  Other Names: ketamine hydrochloride
  Arms: ketamine
Drug: Normal saline — Normal saline will be used for placebo in this group
  Other Names: saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the relative feasibility of 2 potential functional measures of target engagement (Glx MRS, BOLD fMRI) to systematically assess mGluR 2/3 in drug development for psychotic spectrum disorders.

DETAILED DESCRIPTION:
This is a pilot study of healthy subject to assess the feasibility of Glx MRS and BOLD fMRI to measure ketamine induced changes in glutamatergic indices. The investigators will randomize 18 subjects at each site. Subjects will be randomized to ketamine or placebo in a 2:1 ratio and receive two drug challenges separated by at least two weeks. Ketamine challenge is used to induce a "glutamate surge" within prefrontal brain regions that can be detected using neurochemical and functional imaging techniques. Each subject will receive MRS and BOLD fMRI during each challenge day. The goal of the pilot study is to assess the feasibility of both the proposed ketamine challenge paradigm and of the proposed imaging-based biomarkers. Specific indices to be used in assessing feasibility will include effect size, cross-site and cross-subject reliability, safety, and subject tolerability as similar studies will be performed independently at Yale and UC Davis. Second this information will be used to select and refine final study parameters for a subsequent full proof-of-clinical mechanism (POCM) study investigating the effect of Pomaglumetad on ketamine-induced MRS and fMRI effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Negative Urine Toxicology
* No present or past psychiatric conditions (including substance abuse or dependence, with the exception of nicotine dependence)
* No family history of schizophrenia in a first-degree relative

Exclusion Criteria:

* Any current DSM IV Axis I disorder and/or past substance abuse of dependence (nicotine dependence is allowed)
* Any current use of amphetamines, opiates, cocaine, sedative-hypnotics, or cannabis
* Current (i.e., within the last 3 months) treatment with any psychotropic medications
* Pregnancy, lactation, or lack of use of effective birth control
* Presence of positive history of significant medical or neurological illness (including any history of seizure), including high blood pressure (SBP >140, DBP >90), low blood pressure (SBP <100, DBP <60), orthostatic BP change>20% (1/3 SBP + 2/3 DBP) or cardiac illness or resting heart rate >100 or <50
* History of significant violent behavior
* History of recreational ketamine use, recreational PCP use, or an adverse reaction to ketamine. Subjects who have participated prior research ketamine studies will be eligible providing they have participated in no more than 5 previous research ketamine infusions. Subjects can have infusions not more frequently than biweekly and not more than 1/month on average, therefore subjects entering the study will need to wait 1 month if they had a single infusion and 6 weeks if they have had two closely spaced infusions.
* Contraindication to MRI scanning, including metal implants or claustrophobia. Metal implants, pacemaker, other metal (e.g. shrapnel or surgical prostheses) or paramagnetic objects contained within the body which may present a risk to the subject or interfere with the MR scan, as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects", F.G. Shellock, Lippincott Williams and Wilkins NY 2001
* Color Blindness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Lieberman, MD, Principal Investigator — New York State Psychiatric Institute
Locations (3):
- United States (3):
  - University of California Davis, Sacramento, California
  - Yale University, New Haven, Connecticut
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Derived] Javitt DC, Carter CS, Krystal JH, Kantrowitz JT, Girgis RR, Kegeles LS, Ragland JD, Maddock RJ, Lesh TA, Tanase C, Corlett PR, Rothman DL, Mason G, Qiu M, Robinson J, Potter WZ, Carlson M, Wall MM, Choo TH, Grinband J, Lieberman JA. Utility of Imaging-Based Biomarkers for Glutamate-Targeted Drug Development in Psychotic Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Jan 1;75(1):11-19. doi: 10.1001/jamapsychiatry.2017.3572. PMID 29167877

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 65 subjects were randomized, with results (Number started) reported for the 59 subjects randomized subjects with at least one valid scan
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 39 | 20
Completed | 39 (number of subjects with at least one valid scan) | 20 (number of subjects with at least one valid scan)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketamine: randomized to ketamine
- Placebo: randomized to placebo
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 39 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (9.6) | 32.2 (10.2) | 31.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 18 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Glutamate + Glutamine (Glx) Response
Description: Compare changes in Glx response to infusion of ketamine vs placebo, as measured by proton magnetic resonance spectroscopy (¹H MRS). Calculated by post-pre changes in the Glx over creatinine ratios, with higher values indicating higher Glx/creatinine ratios.
Time Frame: Day 1
Population: Glx response in 1st 15 minutes post ketamine
Measure: Mean (Standard Error); unit: Glx over creatinine ratio
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 31 | 16
Glx over creatinine ratio | 0.015 (.002) | 0.007 (.003)

2. Other Pre Specified Outcome: Pharmacological Blood-oxygen-level Dependent (pharmacoBOLD) Response
Description: Compare changes inpharmacoBOLD in response to infusion of ketamine vs. placebo, as measured by resting state functional magnetic resonance imaging. Calculated by post-pre changes, with higher values indicating higher response
Time Frame: Day 14
Measure: Mean (Standard Error); unit: BOLD signal units
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 34 | 19
BOLD signal units | .91 (.1) | -0.27 (0.14)

ADVERSE EVENTS:
Arm/Group | Ketamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/20
Other Adverse Events (participants affected / at risk) | 6/39 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=39) | Placebo (N=20)
ketamine psychological effect (Psychiatric disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No